CLINICAL TRIAL: NCT01199783
Title: Application of Daptomycin in MRSA Infected Diabetic Foot in Comparison to Vancomycin Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient number to be enrolled not reachable in prospected time frame, decision to stop the study prematurely was made.
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Diethelm Tschoepe, Prof. Dr. Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCBC134ADE02T
Record Dates: First submitted 2010-04-29; First posted 2010-09-13 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot,MRSA,; Complicated skin and skin structure infections; Antimicrobial therapy; Daptomycin
MeSH Terms: conditions — Diabetic Foot | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin (Experimental): Infusion of Daptomycin (6 mg/kg bodyweight) once daily
  Interventions: Drug: Daptomycin
- Vancomycin (Active Comparator): Vancomycin once daily (effective blood-plasma concentration of 15 mg/l)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin — Infusion (6 mg/kg/bodyweight) once daily
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Vancomycin — vancomycin once daily (effective blood-plasma concentration of 15 mg/L)
  Arms: Vancomycin

SUMMARY:
Objective of the study is to test whether Daptomycin (6 mg/kg bodyweight) is non-inferior in treatment of severe diabetic foot infections (MRSA) in comparison to antibiotic treatment with Vancomycin (effective blood-plasma concentration of 15 mg/l). In case of microbiologically confirmed gram-negative co-infection effective antibiotic treatment according to microbiologic analysis will be administered upon medical decision in both therapy groups. The study will be carried out as a randomized, open label study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and Type 2 Diabetes mellitus
* MRSA infected foot ulcus Wagner 1-2 without primary surgical intervention
* Therapy duration will last at least more than 5 days
* men and women age 18 - 80 years
* Declaration of patient's consent
* Ability and willingness to give written informed consent and to comply with the requirements of the study
* Sexually active females, unless surgically sterile, must be willing to use 2 forms of contraception through the end of the study. Sexually active woman must, except if they were surgically sterilized, have to use for already 30 days before first dose of study medication an effective method of pregnancy prevention. Acceptable forms of contraception for female subjects include: oral, transdermal, injectable or implanted contraceptives, intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, absolute waiver of sexual intercourse, use of a condom by the sexual partner, or sterile sexual partner. Male subjects with partners of child-bearing potential should use barrier contraception in addition to having their partners use another method of contraception.

Exclusion Criteria:

* Osteomyelitis according to international consensus guideline (3 of 5 criteria apply for diagnosis)
* Presence of a severe nephropathy (creatinine clearance < 30 ml/min)
* Advanced diabetic retinopathy
* Simultaneous participation in another study or participation in a study in the past 30 days
* Non permissible concomitant medication e.g. therapy regimen using several antibiotics
* Contraindication for antibiotics
* Dialysis essential
* Pregnancy (to be determined by pregnancy test) or unsafe contraception
* Neutropenia
* immunosuppression (oral immunosuppressives, Corticoids exaggerating 7.5 mg Prednisolon-equivalents)
* Chronic liver disease (AST or ALT increased to 10fold, bilirubin increased to threefold compared to normal values)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, Prof Dr Dr, Principal Investigator — Herz- und Diabeteszentrum NRW
Locations (1):
- Herz- und Diabeteszentrum, Bad Oeynhausen, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was prematurely stopped after inclusion of 1 patient who was randomized to the Daptomycin arm. During the trial it became obvious that the patient number to be enrolled is not reachable in prospected time frame, thus, the decision to stop the study prematurely was made.
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin
Started | 1 (Only one patient entered the trial and was randomized to the Daptomycin group) | 0
Completed | 1 (study completed, endpoint reached) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: as only one patient was randomized and study was terminated prematurely, no analysis was and will be performed
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (0) |  | 71 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  Germany | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response of the Infection at Test-of-cure (TOC) at Day 14 Post Therapy
Description: Clinical response of the infection at test-of-cure (TOC) at day 14 post therapy by doctoral's decision
  For each of the patients included in the study the clinical outcome at TOC should be assessed using the following criteria:
  Cure: resolution of all clinical signs and symptoms of infection and a healing wound after ≥ 5 days of therapy Improvement: resolution of ≥ 2 - but not all- clinical signs and symptoms of infection after ≥ 5 days of therapy (only used at the end of therapy) Failure: persistence or progression of baseline clinical signs and symptoms of infections after ≥ 2 days of therapy Missing: patients received therapy for less than 2 days Indeterminate: circumstances preclude classification
  Duration of Treatment The duration of treatment will be evaluated as the number of inpatient and outpatient days the patient received antibiotic therapy, even if non-consecutive.
  Time to Clinical Improvement If according to the patient record
Time Frame: 14 days
Population: Participant's infection was solved at day 5 of the study - only 1 participant was treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 1 | 0
Participants | 1 |

2. Secondary Outcome: Duration of Therapy
Description: Duration of therapy until infection was solved in days
Time Frame: 14 days
Population: only one participant was randomized and analyzed
Measure: Number; unit: days
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 1 | 0
days | 5 |

3. Secondary Outcome: Therapy Related Complications
Description: Number of therapy related complications
Time Frame: within time frame of 14 days
Population: only one randomized particpant available for evaluation
Measure: Number; unit: number of events
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 1 | 0
number of events | 0 |

4. Secondary Outcome: Number of Successful Treatments at TOC
Description: * from the clinician point of view (clinical signs and symptoms)
  * from microbiological analysis
Time Frame: within time frame of 14 days
Population: only one participant was randomized and analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 1 | 0
Participants | 1 |

5. Secondary Outcome: Rate of Amputations Due to Infection
Description: Rate of amputations due to infection given as number of events per total events in the study in percent
Time Frame: within time frame of 14 days
Population: only one participant was randomized and analyzed, no amputation occured
Units Other Than Participants: number of amputations
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 1 | 0
Number analyzed (number of amputations) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: only one participant was reandomized to Daptomycin treatment and analyzed, no patients in the comparator group
Arm/Group | Daptomycin | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
recruitment of patients turned out to be limiting in a way that in due time the study could not be performed - therefore the decision to stop the trial was made

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No